CLINICAL TRIAL: NCT05388136
Title: Multicenter Randomized Trial Comparing an Individualized De-intensified and Conventional Follow-up Strategy After Curative Treatment in Head and Neck Cancer
Brief Title: Trial Comparing Different Follow-up Strategies
Acronym: DeintensiF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1685 DeintensiF; SNCTP000005198 (Other: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Cancer
Keywords: Follow up schedule; Patient reported outcomes; Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Conventional (standard) FU entails frequent clinical exams and routine imaging (17 visits including a visit at randomization, plus 4 or 7 imaging depending on smoking habits of the participant) during 5 years of FU.
  PRO with rating scale is to be completed monthly by the participant, but no alert will be generated and the participating center will not arrange urgent appointment, except in case of self-referral for any reasons.
  Interventions: Procedure: Conventional follow up schedule with imaging
- Individualized Deintensified Arm (Experimental): Individualized de-intensified FU entailing less frequent clinical exams and no routine imaging (11 visits including visit at randomization) without any routinely planned imaging during 5 years of FU.
  PRO with rating scale is to be completed monthly by the participant. The PRO result will trigger an alert to the participant and to the site in conditions indicating possible REC/SPM. In case of possible (recurrence or secondary primary malignancy) REC/SPM, an 'open urgent appointment' will be arranged for the participant by the participating centers' team within 2 weeks.
  Interventions: Procedure: Deintensified follow up schedule without imaging

INTERVENTIONS:
Procedure: Conventional follow up schedule with imaging — Frequent of follow up visit and imaging
  Arms: Control Arm
Procedure: Deintensified follow up schedule without imaging — Less intense follow up visit without imaging
  Arms: Individualized Deintensified Arm

SUMMARY:
There is an ongoing debate about the optimal duration, frequency and extent of follow-up (FU) after treatment with curative intent (aimed at complete cure) in patients with head and neck cancer (HNC). The present study aims to answer these questions and thus provide a scientifically sound, evidence-based basis for the current debate. The aim is to develop a more personalized follow-up strategy with patient involvement. The study contains an internal pilot phase and a main phase.

Pilot phase, started in Oct 2022:

Sample size: 20 participants Duration: 2 years (12 months recruitment, 12 months FU) Planned First-Participant-In: Oct 2022 Planned Last-Participant-Out: Oct/2024

Main study, not yet started awaiting for funding :

Sample size: 550 participants Estimated duration: 8 years (recruitment period: 3 years, FU period: 5 years) Planned First-Participant-In: Q4/2023 Planned Last-Participant-Out: Q4/2031

DETAILED DESCRIPTION:
The study will be conducted in a two-arm design, with a control group receiving conventional aftercare and a group receiving less intensive, individualized aftercare. Patients in both groups will be strongly sensitized or trained to the symptoms of cancer recurrence or second tumor. Assignment to one of the two groups is randomized. The study starts with a internal pilot phase of one year aiming to proof the feasibility of recruitment and participant's adherence to the randomized FU scheme. When the pilot phase proved feasibility showed positive result, we will conduct the main study which lasts 5 years for all participants.

For the control group (standard follow-up), medical check-ups are performed at 3-monthly intervals in the first 3 years after completion of therapy, then 4 - 6-monthly until completion of the follow-up period after 5 years. In addition, imaging is scheduled 12 and 24 months after the end of therapy. In addition, imaging examinations (magnetic resonance imaging or computed tomography) are scheduled 6 and 18 months after study inclusion. For active and former smokers, a CT scan of the lungs is scheduled at 30, 42, and 54 months.

In the experimental group (individualized, deintensified follow-up), medical examinations are scheduled only every six months from the beginning and there are no fixed appointments for imaging. In the latter follow-up strategy, the focus is more on the symptoms of the patients.

In the study, participants in both groups document their symptoms monthly in a patient reported-outcome (PRO) questionnaire with possible signs of disease indicating a recurrence of head and neck cancer or a new secondary tumor. For the pilot study, a paper PRO will be used, while in the main study a electronic PRO is planned. In the less intensive, individualized follow-up strategy, the answers to the symptom questionnaires are checked monthly and, depending on the severity and development of the symptoms, a warning is given and a timely follow-up appointment is organized. During this appointment, it will be decided if additional examinations such as imaging and/or tissue sampling are necessary. This means that fewer examinations are not necessarily performed overall, but at times when there is an increased likelihood that a clinically relevant finding will also be found.

Disease progression will be monitored for 5 years.

ELIGIBILITY:
Inclusion criteria

1. Histopathologically proven invasive HNSCC of the oral cavity (except lip), oropharynx, hypopharynx or larynx
2. ≥18 years of age
3. In non-surgically treated HNSCC: clinical/radiological stage II-IV (excluding M1) according to the UICC / TNM 8th ed. In surgically treated HNSCC: pathological stage II-IV (excluding M1) according to the UICC / TNM 8th ed.
4. Treatment with curative intent, regardless of treatment modality (mono- or multimodal), and FU planned at the participating study center.

   Remark: Patients with one synchronous HNSCC of the oral cavity, oropharynx, hypopharynx and larynx, all treated with curative intent and all in complete remission are eligible. Synchronous tumor must have a less advanced stage than the index tumor used for stratification or in case of equal stage, the synchronous tumor must be the tumor with the better prognostic. (Rules: Better to worse prognostic: Larynx > Oropharynx > Oral cavity > Hypopharynx.) The modality of the treatment must be the same as for the index tumor or less intense.
5. Radiological confirmation of complete remission of disease and no SPM from the 3rd to 6th month after treatment for all stages (minimal demanded imaging: head and neck (H&N) MRI or H&N CT scan and CT scan covering chest to pelvis (with contrast if not contraindicated); or preferable whole-body 18FDG-PET/CT or PET/MRI for patients with ≥T3 and/or N+).

   Note: Patients with positive or equivocal imaging/clinical findings are allowed if the tumor is ruled out by multidisciplinary tumor board decision (e.g. as a consequence of biopsy and/or multiple imaging).
6. Clinical confirmation of complete remission of disease through H&N examination including endoscopy of the pharynx and larynx at the time of enrolment, that is 6 months (+/- 4 weeks) after the last HNSCC treatment
7. Agreement for long term FU (5 years) and all visits are to be performed at the participating center
8. Written informed consent, signed by the patient and the investigator

Exclusion Criteria

1. Initial clinical stage I and/or M1 HNSCC (according to the UICC / TNM 8th ed.)
2. Nasopharyngeal cancer and carcinoma of unknown primary
3. Any other previously treated HNC (including parotid and thyroid gland cancer) except for curatively and adequately treated cutaneous carcinoma in-situ, basal cell carcinoma and locally confined T1 squamous cell carcinoma of the skin without any sign of tumor recurrence at the time of screening
4. Any other synchronous malignancy except for one curatively and adequately treated HNSCC of the oral cavity, oropharynx, hypopharynx and larynx, basal cell carcinoma, locally confined T1 squamous cell carcinoma of the skin, low-risk prostate cancer, carcinoma in-situ of the skin or uterine cervix without any sign of tumor recurrence at the time of screening.
5. Any other metachronous malignancy within the last 5 years except for curatively and adequately treated basal cell carcinoma, locally confined T1 squamous cell carcinoma of the skin, low-risk prostate cancer, carcinoma in-situ of the skin or uterine cervix without any sign of tumor recurrence at the time of screening.
6. Participation in another study entailing regular medical exams by ENT specialists or persons involved in the oncological treatment, or regular imaging
7. Pregnant or breastfeeding women
8. Presence of any conditions that potentially hamper compliance with the study protocol and FU schedule at the participating center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2031-10-11 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | Up to 5 years
  Death from any cause is defined as the time interval between the date of randomization and the date of death up to 5 years i.e. patients who are not known to have died will be censored at the date of the last time point at which they were known to be alive (quantified by the 5-year RMST).

SECONDARY OUTCOMES:
Death from head and neck cancer | Up to 5 years
  Time to HNC-specific death
Death from any cancer | Up to 5 years
  Time to cancer-specific death
First biopsy-proven REC or SPM | Up to 5 years
  Based on participating centers' assessment according to the Union for International Cancer Control (UICC)/ tumor, nodes, metastasis (TNM) 8th ed.
General health-related Quality of Life (QoL) | Up to 5 years
  As assessed every 6 months over 5 years by means of the European Organisation for Research and Treatment of Cancer, Core Quality of Life of Cancer Patients (EORTC QLQ-C30)a scale of 1 - 4 are used to assess each condition and a higher scores mean a worse outcome
Head and neck cancer-specific health-related QoL | Up to 5 years
  As assessed every 6 months over 5 years by means of the European Organisation for Research and Treatment of Cancer, Head and Neck Cancer Module (EORTC QLQ-HN43), a scale of 1 - 4 are used to assess each condition and a higher scores mean a worse outcome
Compliance with scheduled follow up assessments | Up to 5 years
  Defined as percentage of scheduled follow up visits attended
Number of regularly scheduled in-person visits | Up to 5 years
Number of in-person visits triggered by the recommendation of the PRO | Up to 5 years
Number of self-referral in-person visits | Up to 5 years
Number of any in-person visits | Up to 5 years
Fear of Recurrence (REC) | Up to 5 years
  Assessed by a rating scale (0 - 4) question within the PRO questionnaire, and a higher scores mean a worse outcome
Head and neck caner-specific healthcare utilization | Up to 5 years
  Defined as any regular and emergency visits to any physician, hospitalizations and treatments for HNC-related reasons

OTHER OUTCOMES:
Type and grading of specific treatment-related adverse events and outcome | Up to 5 years
Characteristics of REC/ secondary primary malignancy (SPM) | Up to 5 years
  Diagnostic modalities that lead to detection of REC/SPM, incidence, site, stage, and whether it is amenable to curatively-intended salvage therapy
Adherence to electronical signs/symptom monitoring and visits that are triggered by the PRO | Up to 5 years
  Defined as the number of PRO questionnaires that were completed and the number of follow up visits that were triggered by the PRO in which the participant attended

CONTACTS AND LOCATIONS:
Overall Officials: Roland Giger, Dr. med., Principal Investigator — Inselspital, University Hospital Bern
Locations (3):
- Switzerland (3):
  - Inselspital, University Hospital Bern, Bern
  - Luzerner Kantonsspital, Klinik für Hals-,Nasen-,Ohren-und Gesichtschirurgie, Lucerne
  - Universitätsspital Zürich, Klinik für Ohren-, Nasen-, Hals- und Gesichtschirurgie, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller M, Visini M, Mueller SA, Stadler T, Rajan GP, Morand GB, Hool SL, Schanne DH, Balermpas P, Limacher A, Chan S, Trelle S, Elicin O, Giger R. DeintensiF: Standard versus individualized deintensified follow-up after curative treatment in head and neck cancer: protocol of a randomized pilot study. Pilot Feasibility Stud. 2025 May 16;11(1):69. doi: 10.1186/s40814-025-01651-3. PMID 40380278